CLINICAL TRIAL: NCT00222573
Title: Clopidogrel Or Metoprolol in Myocardial Infarction Trial
Brief Title: Efficacy and Safety of Adding Clopidogrel to Aspirin or Use of Metoprolol in Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Sanofi (Industry); AstraZeneca (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: COMMIT-CCS2; H6RDCN0
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2006-05-05 (Estimated); Status verified 2005-03

CONDITIONS: Acute Myocardial Infarction
Keywords: clopidogrel; metoprolol; myocardial infarction; randomised trial
MeSH Terms: conditions — Myocardial Infarction | interventions — Clopidogrel; Metoprolol

INTERVENTIONS:
Drug: clopidogrel and metoprolol

SUMMARY:
COMMIT/CCS2 is a large randomised trial of the effects of clopidogrel plus Aspirin versus Aspirin alone in acute heart disease. Patients presenting within 24 hours of the onset of suspected acute MI were potentially eligible provided they were thought to have ST elevation or other ischaemic ECG abnormality with no clear indication for, or contraindication to, trial treatment. All patients were to be given 162 mg ASA daily and, in addition, 75 mg clopidogrel daily or matching placebo for 4 weeks or until prior discharge or death. (Patients were also randomised separately in a 2 X 2 factorial design between metoprolol versus placebo.) The two main study endpoints are death and the composite outcome of death, non-fatal reinfarction or stroke during the scheduled treatment period in hospital.

DETAILED DESCRIPTION:
Clopidogrel

Despite considerable improvements in the emergency treatment of acute myocardial infarction (MI), including the use of aspirin, early mortality and morbidity remain high. The antiplatelet agent clopidogrel adds to the benefit of aspirin in acute coronary syndromes without ST-segment elevation, but its effects on mortality and morbidity in patients with ST-elevation MI were unclear.

45,852 patients admitted to 1250 hospitals within 24 hours of the onset of suspected acute MI were randomly allocated to receive clopidogrel 75 mg daily or matching placebo (both in addition to aspirin 162 mg daily). 93% had ST-segment elevation or bundle branch block, and 7% had ST-segment depression. Treatment was to continue until discharge or up to a maximum of 4 weeks in hospital (mean 15 days in survivors), and 93% completed it. The two pre-specified co-primary outcomes were: (i) the composite of death, reinfarction or stroke; and (ii) death from any cause during the scheduled treatment period. Comparisons were between all clopidogrel-allocated and all placebo-allocated patients (ie, "intention-to-treat"), and used the log-rank method.

Allocation to clopidogrel produced a highly significant 9% (95% CI 3-14) proportional reduction in the primary composite outcome of death, reinfarction or stroke (2121 [9.2%] clopidogrel vs 2310 [10.1%] placebo; p=0.002), corresponding to 9 (SE 3) fewer events per 1000 patients treated for about 2 weeks. There was also a significant 7% (95% CI 1-13) proportional reduction in the co-primary outcome of any death (1726 [7.5%] vs 1845 [8.1%]; p=0.03). These effects on death, reinfarction and stroke appeared to be consistent across a wide range of patients and independent of other treatments being used. Considering all transfused, fatal or cerebral bleeds together, no significant excess risk was observed with clopidogrel, either overall (134 [0.58%] vs 125 [0.55%]; p=0.59), or among patients aged 70 years or older (50 [0.84%] vs 43 [0.72%]; p=0.48) or among those given fibrinolytic therapy (74 [0.65%] vs 72 [0.63%]; p=0.88).

In a wide range of patients with acute MI, adding clopidogrel 75 mg daily to aspirin and other standard treatments (such as fibrinolytic therapy) reduces mortality and major vascular events in hospital, without any material increase in major bleeding.

Metoprolol

Despite previous randomised trials of early beta-blocker therapy in the emergency treatment of suspected acute myocardial infarction (MI), substantial uncertainty has persisted about the value of adding it to currently standard interventions (eg, aspirin and fibrinolytic therapy), and the balance of potential benefits and hazards was unclear even in high-risk patients.

45852 patients admitted to 1250 hospitals within 24 hours of the onset of suspected acute MI were randomly allocated to receive metoprolol (up to 15 mg intravenous followed by 200 mg oral daily) or matching placebo. 93% had ST-segment elevation or bundle branch block, and 7% had ST-segment depression. Treatment was to continue until discharge or up to a maximum of 4 weeks in hospital (mean 15 days in survivors), and 89% completed it. The two pre-specified co-primary outcomes were: (i) the composite of death, reinfarction or cardiac arrest; and (ii) death from any cause during the scheduled treatment period. Comparisons were between all metoprolol-allocated and all placebo-allocated patients (ie, "intention-to-treat"), and used the log-rank method.

Neither of the co-primary outcomes was significantly reduced by allocation to metoprolol. For the primary composite outcome of death, reinfarction, or cardiac arrest, 2166 (9.4%) patients had at least one such event among the 22 929 allocated metoprolol compared with 2261 (9.9%) among the 22 923 allocated matching placebo (odds ratio [OR] 0.96 [95% CI 0.90-1.01]; p=0.1). For the co-primary outcome of death alone, there were 1774 (7.7%) in the metoprolol group versus 1797 (7.8%) in the placebo group (OR 0.99 [0.92-1.05]; p=0.69). Allocation to metoprolol was associated with 5 fewer people having reinfarction (464 [2.0%] metoprolol vs 568 [2.5%] placebo; OR 0.82 [0.72-0.92]; p=0.001) and 5 fewer having ventricular fibrillation (581 [2.5%] vs 698 [3.0%]; OR 0.83 [0.75-0.93]; p=0.001) per 1000 treated. Overall, these reductions were counter-balanced by 11 more per 1000 allocated metoprolol developing cardiogenic shock (1141 [5.0%] vs 885 [3.9%]; OR 1.30 [1.19-1.41]; p<0.00001). The excess of cardiogenic shock was chiefly during days 0-1 after hospitalisation, whereas the reductions in reinfarction and ventricular fibrillation emerged more gradually. Consequently, the overall effect on death, reinfarction, arrest or shock was significantly adverse during days 0-1 and significantly beneficial thereafter. There was substantial net hazard among haemodynamically unstable patients and moderate net benefit among those who were relatively stable, particularly after days 0-1.

The use of early beta-blocker therapy in acute MI reduces the risks of reinfarction and ventricular fibrillation, but increases the risk of cardiogenic shock, especially during the first day or so after hospitalisation. Consequently, it may generally be prudent to consider starting beta-blocker therapy in hospital only when the haemodynamic condition following MI has stabilized (and then, based on previous evidence, to continue such therapy long-term following discharge).

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with ST elevation, left bundle branch block or ST depression within 24 hours of the onset of the symptoms of suspected acute MI

Exclusion Criteria:

* clear indications for, or contraindications to, any of the study treatments

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46000
Dates: Start 1999-07; Study Completion 2005-02

PRIMARY OUTCOMES:
Death and the composite outcome of death, non-fatal reinfarction or stroke

SECONDARY OUTCOMES:
Major cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Rory Collins, Msc, Study Chair — University of Oxford; Lisheng Liu, MD, Study Chair — Institute of cardiovascular diseases, Fuwai hospital, Chinese academy of medical sciences
Locations (2):
- Institute of Cadiovascular diseases, Fuwai hospital, Chinese academy of medical sciences, Beijing, China
- Clinical Trial Service Unit and Epidemiological Studies Unit, Oxford, United Kingdom

REFERENCES:
- [Result] Chen ZM, Pan HC, Chen YP, Peto R, Collins R, Jiang LX, Xie JX, Liu LS; COMMIT (ClOpidogrel and Metoprolol in Myocardial Infarction Trial) collaborative group. Early intravenous then oral metoprolol in 45,852 patients with acute myocardial infarction: randomised placebo-controlled trial. Lancet. 2005 Nov 5;366(9497):1622-32. doi: 10.1016/S0140-6736(05)67661-1. PMID 16271643
- [Result] Hubner G, Golbik R, Meshalkina LE. A method for determination of transketolase activity based on the use of a pH indicator. Biochem Int. 1992 Mar;26(3):545-50. PMID 1627164
- [Derived] Steingrimsson JA, Hanley DF, Rosenblum M. Improving precision by adjusting for prognostic baseline variables in randomized trials with binary outcomes, without regression model assumptions. Contemp Clin Trials. 2017 Mar;54:18-24. doi: 10.1016/j.cct.2016.12.026. Epub 2017 Jan 4. PMID 28064029
- [Derived] Chen ZM, Jiang LX, Chen YP, Xie JX, Pan HC, Peto R, Collins R, Liu LS; COMMIT (ClOpidogrel and Metoprolol in Myocardial Infarction Trial) collaborative group. Addition of clopidogrel to aspirin in 45,852 patients with acute myocardial infarction: randomised placebo-controlled trial. Lancet. 2005 Nov 5;366(9497):1607-21. doi: 10.1016/S0140-6736(05)67660-X. PMID 16271642
- See also: study website — http://www.commit-ccs2.org